CLINICAL TRIAL: NCT01820611
Title: Arcos Revision Stem: Evaluation of Clinical Performance
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: GBMET.CR.US19
Record Dates: First submitted 2013-03-19; First posted 2013-03-29 (Estimated); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Deformity; Fracture; Complications; Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Congenital Abnormalities; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- With Bonemaster HA: 100 patients using Arcos Revision Stem System with BoneMaster Hydroxyapatite
  Interventions: Device: Arcos Revision Stem System

INTERVENTIONS:
Device: Arcos Revision Stem System — Revision Hip System

SUMMARY:
The primary purpose of this study is to evaluate the clinical performance of the Arcos Revision Stem system, determine the stability of the implants, and evaluate any relationship between Paprosky bone defect level and the success of the Arcos Stem.

DETAILED DESCRIPTION:
Primary Endpoint: survivorship and revision rate up to 5 years post-operatively Secondary Endpoints: Stability and Fixation of Arcos Hip by radiographic assessment, Relationship between bone defect level and survivorship, Oxford Hip Score and Harris Hip Score post-operative, Adverse events, complications.

Case Report Forms: Demographic Data, Paprosky Acetabular/Femoral Defects, Operative Data, Oxford Hip Score, Harris Hip Score, Collection of X-rays, Radiographic Evaluation form, Adverse Events, Revisions, Lost to Follow-up, and Protocol Deviations

200 patients: 100 with BoneMaster HA, 100 without BoneMaster HA. Up to 10 sites globally will be used to fulfill enrollment in this study.

All cases enrolled will be those implanted with either the Cone, Broached, or Calcar Proximal Body and one of the five distal options (Slotted, Bullet-tip, Interlocking, STS, or ETO).

To be included in the study, a patient must have received a revision total hip arthroplasty with the Arcos system. The Arcos system is to be used in accordance to the indications for use and contraindications detailed in the approved labeling of the device.

Study time perspective:

Collection of retrospective data in supplement to the data collected in the course of the prospective study to compensate total enrolment goal. This is applicable for 3 sites: Finland, United Kingdom (NHS Sheffield), Spain.

All patients enrolled in the study will be followed up as to the same time points for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid arthritis
* Correction of functional deformity
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable using other techniques.
* Revision of previously failed total hip arthroplasty.

The Arcos™ Modular Femoral Revision System hip components are single-use implants, intended for uncemented use only.

Only subjects who have received or have already been scheduled to receive hip surgery with the Arcos Revision Stem System will be included in this outcomes study.

Additional Inclusion Criteria:

* No age limit, however, the patient must have reached full skeletal maturity.
* Willing to return for follow up evaluation.

Exclusion Criteria:

Absolute contraindications include: active infection, sepsis, and osteomyelitis.

Relative contraindications include:

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, or neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who had a revision to a total hip replacement using the Arcos Revision Stem Hip System.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2013-02; Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (5):
- Turku University Hospital, Turku, Finland
- Hospital Universitari Mutua, Barcelona, Spain
- Uddevalla Hospital, Uddevalla, Sweden
- United Kingdom (2):
  - Hinchingbrooke Hosptial, Cambridge
  - NHS - Sheffield Teaching Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 74 cases who received the Arcos hip stem were evaluated at 5 study centers in Europe.
Pre-assignment Details: After checking the operative records for the prospective and retrospectively enrolled cases, only 74 cases were eligible to be included in the study.
Period: Overall Study
Arm/Group | With Bonemaster HA
Started | 74
Completed | 56
Not Completed | 18
Not completed — Death | 8
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Population: 74 cases who were eligible to be included in the study.
Groups:
- With Bonemaster HA: Patients using Arcos Revision Stem System with BoneMaster Hydroxyapatite
  Arcos Revision Stem System: Revision Hip System
Arm/Group | With Bonemaster HA
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 19
  Finland | 15
  United Kingdom | 22
  Spain | 18
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.2 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Survivorship
Description: The primary endpoint for this study was implant survival at 5 years post surgery and is presented by the number of cases with the implants unrevised
Time Frame: 5 year post surgery
Population: All study patients
Measure: Count of Participants; unit: Participants
Arm/Group | With Bonemaster HA
Number analyzed (Participants) | 74
Participants | 74

2. Secondary Outcome: Radiographic Evaluation
Description: This outcome measure was to evaluate the stability and fixation of the Arcos hip stem. This was done through radiographic measurements of stability and fixation, outcome, incidence of radiolucencies around the stem. Acetabular radiolucency was also assessed.
Time Frame: 6 weeks, 1 year, 3 years and 5 years Post Surgery
Population: Acetabular and femoral radiolucency was analysed for all study patients for different zones at the outcome measure time frames listed above. The numbers listed below in the count of participants is the number of cases where radiolucency was seen on their X-ray images in different zones and at different follow up time points.
Measure: Count of Participants; unit: Participants
Arm/Group | With Bonemaster HA
Number analyzed (Participants) | 74
Participants
  Number of patients with Acetabular Radiolucency seen in their Xray images, 6 Weeks Zone 1: number analyzed (Participants) | 43
  Number of patients with Acetabular Radiolucency seen in their Xray images, 6 Weeks Zone 1 | 9
  Acetabular Radiolucency, 6 Weeks Zone 2: number analyzed (Participants) | 42
  Acetabular Radiolucency, 6 Weeks Zone 2 | 4
  Acetabular Radiolucency, 6 Weeks Zone 3: number analyzed (Participants) | 43
  Acetabular Radiolucency, 6 Weeks Zone 3 | 1
  Acetabular Radiolucency, 1 Year Zone 1: number analyzed (Participants) | 66
  Acetabular Radiolucency, 1 Year Zone 1 | 12
  Acetabular Radiolucency, 1 Year Zone 2: number analyzed (Participants) | 65
  Acetabular Radiolucency, 1 Year Zone 2 | 5
  Acetabular Radiolucency, 1 Year Zone 3: number analyzed (Participants) | 66
  Acetabular Radiolucency, 1 Year Zone 3 | 8
  Acetabular Radiolucency, 3 Year Zone 1: number analyzed (Participants) | 61
  Acetabular Radiolucency, 3 Year Zone 1 | 13
  Acetabular Radiolucency, 3 Year Zone 2: number analyzed (Participants) | 60
  Acetabular Radiolucency, 3 Year Zone 2 | 4
  Acetabular Radiolucency, 3 Year Zone 3: number analyzed (Participants) | 61
  Acetabular Radiolucency, 3 Year Zone 3 | 7
  Acetabular Radiolucency, 5 Year Zone 1: number analyzed (Participants) | 52
  Acetabular Radiolucency, 5 Year Zone 1 | 10
  Acetabular Radiolucency, 5 Year Zone 2: number analyzed (Participants) | 51
  Acetabular Radiolucency, 5 Year Zone 2 | 4
  Acetabular Radiolucency, 5 Year Zone 3: number analyzed (Participants) | 52
  Acetabular Radiolucency, 5 Year Zone 3 | 7
  Femoral AP View Radiolucency, 6 Weeks Zone 1: number analyzed (Participants) | 41
  Femoral AP View Radiolucency, 6 Weeks Zone 1 | 6
  Femoral AP View Radiolucency, 6 Weeks Zone 2: number analyzed (Participants) | 43
  Femoral AP View Radiolucency, 6 Weeks Zone 2 | 10
  Femoral AP View Radiolucency, 6 Weeks Zone 3: number analyzed (Participants) | 43
  Femoral AP View Radiolucency, 6 Weeks Zone 3 | 4
  Femoral AP View Radiolucency, 6 Weeks Zone 5: number analyzed (Participants) | 43
  Femoral AP View Radiolucency, 6 Weeks Zone 5 | 4
  Femoral AP View Radiolucency, 6 Weeks Zone 6: number analyzed (Participants) | 43
  Femoral AP View Radiolucency, 6 Weeks Zone 6 | 7
  Femoral AP View Radiolucency, 6 Weeks Zone 7: number analyzed (Participants) | 43
  Femoral AP View Radiolucency, 6 Weeks Zone 7 | 9
  Femoral AP View Radiolucency, 1 Year Zone 1: number analyzed (Participants) | 65
  Femoral AP View Radiolucency, 1 Year Zone 1 | 14
  Femoral AP View Radiolucency, 1 Year Zone 2: number analyzed (Participants) | 66
  Femoral AP View Radiolucency, 1 Year Zone 2 | 9
  Femoral AP View Radiolucency, 1 Year Zone 3: number analyzed (Participants) | 66
  Femoral AP View Radiolucency, 1 Year Zone 3 | 6
  Femoral AP View Radiolucency, 1 Year Zone 4: number analyzed (Participants) | 66
  Femoral AP View Radiolucency, 1 Year Zone 4 | 1
  Femoral AP View Radiolucency, 1 Year Zone 5: number analyzed (Participants) | 66
  Femoral AP View Radiolucency, 1 Year Zone 5 | 2
  Femoral AP View Radiolucency, 1 Year Zone 6: number analyzed (Participants) | 65
  Femoral AP View Radiolucency, 1 Year Zone 6 | 7
  Femoral AP View Radiolucency, 1 Year Zone 7: number analyzed (Participants) | 61
  Femoral AP View Radiolucency, 1 Year Zone 7 | 11
  Femoral AP View Radiolucency, 3 Years Zone 1: number analyzed (Participants) | 61
  Femoral AP View Radiolucency, 3 Years Zone 1 | 16
  Femoral AP View Radiolucency, 3 Years Zone 2: number analyzed (Participants) | 62
  Femoral AP View Radiolucency, 3 Years Zone 2 | 5
  Femoral AP View Radiolucency, 3 Years Zone 3: number analyzed (Participants) | 62
  Femoral AP View Radiolucency, 3 Years Zone 3 | 3
  Femoral AP View Radiolucency, 3 Years Zone 5: number analyzed (Participants) | 61
  Femoral AP View Radiolucency, 3 Years Zone 5 | 6
  Femoral AP View Radiolucency, 3 Years Zone 6: number analyzed (Participants) | 61
  Femoral AP View Radiolucency, 3 Years Zone 6 | 7
  Femoral AP View Radiolucency, 3 Years Zone 7: number analyzed (Participants) | 57
  Femoral AP View Radiolucency, 3 Years Zone 7 | 13
  Femoral AP View Radiolucency, 5 Years Zone 1: number analyzed (Participants) | 52
  Femoral AP View Radiolucency, 5 Years Zone 1 | 9
  Femoral AP View Radiolucency, 5 Years Zone 2: number analyzed (Participants) | 53
  Femoral AP View Radiolucency, 5 Years Zone 2 | 4
  Femoral AP View Radiolucency, 5 Years Zone 3: number analyzed (Participants) | 53
  Femoral AP View Radiolucency, 5 Years Zone 3 | 3
  Femoral AP View Radiolucency, 5 Years Zone 5: number analyzed (Participants) | 53
  Femoral AP View Radiolucency, 5 Years Zone 5 | 0.0
  Femoral AP View Radiolucency, 5 Years Zone 6: number analyzed (Participants) | 52
  Femoral AP View Radiolucency, 5 Years Zone 6 | 2
  Femoral AP View Radiolucency, 5 Years Zone 7: number analyzed (Participants) | 49
  Femoral AP View Radiolucency, 5 Years Zone 7 | 7
  Femoral Lateral View Radiolucency, 6 Weeks Zone 8: number analyzed (Participants) | 42
  Femoral Lateral View Radiolucency, 6 Weeks Zone 8 | 12
  Femoral Lateral View Radiolucency, 6 Weeks Zone 9: number analyzed (Participants) | 43
  Femoral Lateral View Radiolucency, 6 Weeks Zone 9 | 9
  Femoral Lateral View Radiolucency, 6 Weeks Zone 10: number analyzed (Participants) | 43
  Femoral Lateral View Radiolucency, 6 Weeks Zone 10 | 3
  Femoral Lateral View Radiolucency, 6 Weeks Zone 12: number analyzed (Participants) | 43
  Femoral Lateral View Radiolucency, 6 Weeks Zone 12 | 3
  Femoral Lateral View Radiolucency, 6 Weeks Zone 13: number analyzed (Participants) | 43
  Femoral Lateral View Radiolucency, 6 Weeks Zone 13 | 7
  Femoral Lateral View Radiolucency, 6 Weeks Zone 14: number analyzed (Participants) | 42
  Femoral Lateral View Radiolucency, 6 Weeks Zone 14 | 6
  Femoral Lateral View Radiolucency, 1 Year Zone 8: number analyzed (Participants) | 64
  Femoral Lateral View Radiolucency, 1 Year Zone 8 | 19
  Femoral Lateral View Radiolucency, 1 Year Zone 9: number analyzed (Participants) | 64
  Femoral Lateral View Radiolucency, 1 Year Zone 9 | 9
  Femoral Lateral View Radiolucency, 1 Year Zone 10: number analyzed (Participants) | 66
  Femoral Lateral View Radiolucency, 1 Year Zone 10 | 4
  Femoral Lateral View Radiolucency, 1 Year Zone 11: number analyzed (Participants) | 66
  Femoral Lateral View Radiolucency, 1 Year Zone 11 | 1
  Femoral Lateral View Radiolucency, 1 Year Zone 12: number analyzed (Participants) | 66
  Femoral Lateral View Radiolucency, 1 Year Zone 12 | 3
  Femoral Lateral View Radiolucency, 1 Year Zone 13: number analyzed (Participants) | 65
  Femoral Lateral View Radiolucency, 1 Year Zone 13 | 10
  Femoral Lateral View Radiolucency, 1 Year Zone 14: number analyzed (Participants) | 62
  Femoral Lateral View Radiolucency, 1 Year Zone 14 | 9
  Femoral Lateral View Radiolucency, 3 Years Zone 8: number analyzed (Participants) | 57
  Femoral Lateral View Radiolucency, 3 Years Zone 8 | 12
  Femoral Lateral View Radiolucency, 3 Years Zone 9: number analyzed (Participants) | 59
  Femoral Lateral View Radiolucency, 3 Years Zone 9 | 7
  Femoral Lateral View Radiolucency, 3 Years Zone 10: number analyzed (Participants) | 59
  Femoral Lateral View Radiolucency, 3 Years Zone 10 | 5
  Femoral Lateral View Radiolucency, 3 Years Zone 12: number analyzed (Participants) | 59
  Femoral Lateral View Radiolucency, 3 Years Zone 12 | 4
  Femoral Lateral View Radiolucency, 3 Years Zone 13: number analyzed (Participants) | 58
  Femoral Lateral View Radiolucency, 3 Years Zone 13 | 7
  Femoral Lateral View Radiolucency, 3 Years Zone 14: number analyzed (Participants) | 55
  Femoral Lateral View Radiolucency, 3 Years Zone 14 | 8
  Femoral Lateral View Radiolucency, 5 Years Zone 8: number analyzed (Participants) | 49
  Femoral Lateral View Radiolucency, 5 Years Zone 8 | 10
  Femoral Lateral View Radiolucency, 5 Years Zone 9: number analyzed (Participants) | 50
  Femoral Lateral View Radiolucency, 5 Years Zone 9 | 3
  Femoral Lateral View Radiolucency, 5 Years Zone 10: number analyzed (Participants) | 50
  Femoral Lateral View Radiolucency, 5 Years Zone 10 | 1
  Femoral Lateral View Radiolucency, 5 Years Zone 12: number analyzed (Participants) | 50
  Femoral Lateral View Radiolucency, 5 Years Zone 12 | 2
  Femoral Lateral View Radiolucency, 5 Years Zone 13: number analyzed (Participants) | 49
  Femoral Lateral View Radiolucency, 5 Years Zone 13 | 3
  Femoral Lateral View Radiolucency, 5 Years Zone 14: number analyzed (Participants) | 48
  Femoral Lateral View Radiolucency, 5 Years Zone 14 | 4

3. Secondary Outcome: EQ5D
Description: The EuroQol 5 Dimension (EQ-5D) is a standardized Instrument widely used to measure health status. It is a self reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes 5 questions referring to mobility, selfcare, daily activities, pain/discomfort, and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. The EQ-5D-5L score ranges from -0.59 to 1, where 1 is the best possible health state. The Visual Analogue Scale (VAS) is a vertical scale ranges from 100 ('The best health you can imagine') to 0 ('The worst health you can imagine') where the patient reports his/her self-rated health.
Time Frame: Preop, 6 Weeks, 1 Year, 3 Years and 5 Years post surgery
Population: All study patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With Bonemaster HA
Number analyzed (Participants) | 74
score on a scale
  Preop EQ-5D: number analyzed (Participants) | 44
  Preop EQ-5D | 0.3 (0.4)
  6 Weeks EQ-5D: number analyzed (Participants) | 43
  6 Weeks EQ-5D | 0.6 (0.2)
  1 Year EQ-5D: number analyzed (Participants) | 46
  1 Year EQ-5D | 0.7 (0.3)
  3 Years EQ-5D: number analyzed (Participants) | 50
  3 Years EQ-5D | 0.7 (0.3)
  5 Years EQ-5D: number analyzed (Participants) | 45
  5 Years EQ-5D | 0.8 (0.2)

4. Secondary Outcome: Oxford Hip Score
Description: The Oxford Hip Score (OHS) is a patient-reported outcome measure that was developed to specifically assess the patient's perspective of outcome following THA. The OHS consists of twelve questions covering function and pain associated with the hip. To calculate the total score, each response is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The Score ranges from 0 - 100 and the outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27.
Time Frame: Preop, 6 weeks, 1 year, 3 years and 5 years post surgery
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With Bonemaster HA
Number analyzed (Participants) | 74
score on a scale
  Preop Oxford Hip Score: number analyzed (Participants) | 44
  Preop Oxford Hip Score | 18.8 (8.6)
  6 Weeks Oxford Hip Score: number analyzed (Participants) | 43
  6 Weeks Oxford Hip Score | 28.3 (8.8)
  1 Year Oxford Hip Score: number analyzed (Participants) | 57
  1 Year Oxford Hip Score | 34.4 (10.9)
  3 Years Oxford Hip Score: number analyzed (Participants) | 62
  3 Years Oxford Hip Score | 36.9 (10.5)
  5 Years Oxford Hip Score: number analyzed (Participants) | 55
  5 Years Oxford Hip Score | 39.3 (8.6)

5. Secondary Outcome: Harris Hip Score
Description: The Harris hip Score (HHS) is an outcome measure that includes a series of questions answered by the patient and physical examinations recorded by a qualified health care Professional. The HHS covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence of deformity (one item, 0-4 points) and range of motion (one item, 0-5 points). The total score can vary from a range of 0 - 100. The outcome score can be categorized as Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70.
Time Frame: Preop, 6 Weeks, 1 Year, 3 Years and 5 Years post surgery
Population: All study patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With Bonemaster HA
Number analyzed (Participants) | 74
score on a scale
  Preop Harris Hip Score: number analyzed (Participants) | 44
  Preop Harris Hip Score | 41.3 (15.6)
  6 Weeks Harris Hip Score: number analyzed (Participants) | 43
  6 Weeks Harris Hip Score | 60.0 (15.3)
  1 Year Harris Hip Score: number analyzed (Participants) | 57
  1 Year Harris Hip Score | 73.0 (21.3)
  3 Years Harris Hip Score: number analyzed (Participants) | 61
  3 Years Harris Hip Score | 78.3 (19.1)
  5 Years Harris Hip Score: number analyzed (Participants) | 52
  5 Years Harris Hip Score | 79.8 (16.8)

ADVERSE EVENTS:
Time Frame: Operative, 6 Weeks, 1 Year, 3 Years and 5 Years
Arm/Group | With Bonemaster HA
All-Cause Mortality (participants affected / at risk) | 8/74
Serious Adverse Events (participants affected / at risk) | 28/74
Other Adverse Events (participants affected / at risk) | 13/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | With Bonemaster HA (N=74)
Deep Infection (Musculoskeletal and connective tissue disorders) | 3 (4) — Deep infection < 6 weeks
Dislocation and Sublaxation (Musculoskeletal and connective tissue disorders) | 3 (5) — Dislocation
Femoral Pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Femoral Pain
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) — Fracture of femoral shaft and trochanter
Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) — Hematoma
Instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Nerve and vascular deficit (Musculoskeletal and connective tissue disorders) | 2 (2) — Nerve and vascular deficit
Superficial Infection (Musculoskeletal and connective tissue disorders) | 1 (1) — Superficial Infection
Wound Drainage and Dehiscence (Musculoskeletal and connective tissue disorders) | 5 (5) — Wound Drainage and Dehiscence
Other Hip Related Adverse Events (Musculoskeletal and connective tissue disorders) | 12 (20) — Pain, trochanteric bolt loosening, contralateral hip surgery, leg reddening, hip athrosis, wound secretion
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | With Bonemaster HA (N=74)
General Complications (Infections and infestations) | 9 (9) — Respiratory infection, Urinary tract infection and infection
General Complications (Nervous system disorders) | 4 (4) — Nerve injury and stroke

LIMITATIONS AND CAVEATS:
The study was initially set up to collect data within two study arms (100 with BoneMaster HA and 100 without BoneMaster HA) globally including up to ten sites. However, the study only ended up enrolling 74 cases with BoneMaster in EMEA across 5 study sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT01820611/Prot_SAP_000.pdf